CLINICAL TRIAL: NCT02383329
Title: Effects of Oral Nutrition Supplements in Children With Disease Associated Underweight
Acronym: MIntS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Michael Chourdakis (Other)
Collaborators: Children's Hospital Zagreb (Other); Universitair Ziekenhuis Brussel (Other); General Hospital Of Thessaloniki Ippokratio (Other); Medical University of Warsaw (Other); Russian Medical Academy of Postgraduate Education (Other); Oxford University Hospitals NHS Trust (Other); Dokuz Eylul University (Other); Ludwig-Maximilians - University of Munich (Other); Aghia Sophia Children's Hospital of Athens (Other); Hacettepe University (Other); Children's Memorial Health Institute, Poland (Other); University Hospital, Lille (Other); Oslo University Hospital (Other); University Hospital, Tours (Other)
Responsible Party: Sponsor-Investigator, Dr. Michael Chourdakis, Lecturer of Medical Nutrition, Aristotle University Of Thessaloniki
Organization: Aristotle University Of Thessaloniki (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AUTh112Med
Record Dates: First submitted 2015-03-02; First posted 2015-03-09 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Disease Associated Underweight
Keywords: malnutrition; Underweight; Oral Nutrition Supplements; Children
MeSH Terms: conditions — Malnutrition; Thinness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Nutritional Supplement (ONS) (Experimental): Diet consultation for the child/family + ONS
  Interventions: Dietary Supplement: The ONS provided to the children intervention group will be a ready to drink age adapted oral nutrition supplement providing 1,5 kcal/ml
- No Oran Nutritional Supplement (ONS) (No Intervention): Diet consultation for the child/family

INTERVENTIONS:
Dietary Supplement: The ONS provided to the children intervention group will be a ready to drink age adapted oral nutrition supplement providing 1,5 kcal/ml — The ONS provided to the children intervention group will be a ready to drink age adapted oral nutrition supplement providing 1,5 kcal/ml
  Arms: Oral Nutritional Supplement (ONS)

SUMMARY:
The purpose of this study is to test whether the provision of ONS to malnourished children across Europe, in addition to standard counselling, will improve weight gain and other outcomes.

The hypothesis to be tested is:

• Supplementation with ONS in malnourished paediatric patients will lead to increased WFH gain, as well as less malnutrition related complications (e.g. infections).

Primary outcome • The change in BMI z-score over the intervention period of 3 months

Secondary outcomes

• The change in WFH-weight for height (z-scores) over the intervention period of 3 months

ELIGIBILITY:
Inclusion Criteria:

1. Children treated at the participating paediatric centres during the study period (inpatients or outpatients)
2. Age between 24 months to 12 years at inclusion
3. WFH at inclusion <- 1,5 SD - >-2,5 SD (based on WHO) OR Decrease in WFH z-score of ≥1 SD within the last 3 months, and underlying disease with high risk of undernutrition
4. Children who would be considered candidates for oral nutrition intervention (but do not need tube feeding)
5. Written informed consent of parents/caregivers

Exclusion Criteria:

1. Children in need of intensive care
2. Inability to consume ONS (e.g. major gastrointestinal dysfunction)
3. Children, for whom normal nutrition intervention would be inappropriate (e.g. food intolerance, allergy)
4. Use of parenteral feeding and/or enteral tube-feeding
5. Severe edema (>0.5 cm pitting edema on the dorsum of the foot)
6. Participation in another intervention study involving investigational or marketed products concomitantly or within two weeks prior to entry into the trial.
7. Children having received enteral nutrition treatment for underweight in the previous month
8. Oncology patients during chemo-, radio-therapy
9. Expected hospital stay at inclusion longer than 7 days

   -

Ages: 24 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 224 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
BMI z-score | 3 months
  The change in BMI z-score over the intervention period of 3 months

SECONDARY OUTCOMES:
Weight change | 3 months
  The change in WFH-weight for height (z-scores) over the intervention period of 3 months
Infectious complications | 3 months
  Frequency of infectious complications (number of days with temperature >38,5°C, number of infections requiring antibiotic use)
Hospital admissions | 3 months
  Admission for hospital inpatient treatments (number of days of hospital stay, number of admissions)
Gastrointestinal complications | 3 months
  Frequency of gastrointestinal complications (number of days with diarrhoea/vomiting as reported by carers). Other GI symptoms could be recorded, as potential reason for lower food intake

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chourdakis, MD PhD, Principal Investigator — AUTH
Locations (19):
- UZ Brussel, Brussels, Belgium
- Children's Hospital Zagreb, Zagreb, Croatia
- France (2):
  - Hospital Jeanne de Flandre, Pediatrics Department, CHRU, Lille
  - CHU Tours, Tours
- Greece (4):
  - Agia Sofia Children's Hospital, Athens
  - Aristotle University of Thessaloniki, School of Medicine, Thessaloniki
  - 1st Paediatric Dept, Hippokration Hospital, AUTH, Thessaloniki
  - 3rd Paediatric Dept, Hippokration Hospital, AUTH, Thessaloniki
- Iran (2):
  - Tehran University of Medical Sciences Tehrān, Children Medical Center, Tehran
  - Mofid Children Hospital, Tehran
- Department of Pediatrics, Women and Children's Division, Oslo University Hospital, Oslo, Norway
- Poland (2):
  - Medical University of Warsaw, Warsaw
  - The Children's Memorial Health Institute, Warsaw
- Russia (2):
  - Kazan State Medical University, Kazan', Tatarstan Republic
  - Russian Medical Academy of Postgraduate Education, Moscow
- Turkey (Türkiye) (4):
  - Dokuz Eylul University,, Izmir, Inciralti-izmir
  - Hacettepe University, Ankara, Ankara
  - Ankara University School of Medicine, Ankara
  - Inönü University School of Medicine, İnönü